CLINICAL TRIAL: NCT05484804
Title: Reducing Racial Disparities in Maternal Care Through Data-Based Accountability and Doula Support
Brief Title: Accountability for Care Through Undoing Racism & Equity for Moms
Acronym: ACURE4Moms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); UNC Health Foundation (Unknown); The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1541
Record Dates: First submitted 2022-07-22; First posted 2022-08-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Maternal Health; Maternal Mortality; Low Birthweight; Racism; Implicit Bias
MeSH Terms: conditions — Maternal Death; Racism; Bias, Implicit | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Arm 1 (Standard Care): NC Medicaid Care Management Arm 2 (Data Accountability and Transparency): NC Medicaid Care Management + Practice-level Data Accountability interventions Arm 3 (Community-Based Doula Support): NC Medicaid Care Management + CBD support intervention for high-risk women during pregnancy and postpartum Arm 4 (Data Accountability and Transparency + Community-Based Doula Support): NC Medicaid Care Management + both Arm 2 and Arm 3 interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard Care (No Intervention): Pregnant patients with Medicaid insurance are screened for risk factors for low birthweight, and high-risk patients receive intensive care management.
- Data Accountability and Transparency (Active Comparator): Pregnant patients with Medicaid insurance are screened for risk factors for low birthweight, and high-risk patients receive intensive care management. Additionally, practices receive 2 additional patient-level interventions, including: 1) Support from a Practice Facilitator to help implement the interventions and build workflows and quality improvement cycles; 2) Use of a Maternal Warning System for missed visits, elevated blood pressures, and prenatal aspirin eligibility; 3) Use of a Data Dashboard that displays outcome data stratified by race, ethnicity, age, and preferred language; and 4) Maternal Health Equity Education & Training sessions.
  Interventions: Other: Data Accountability and Transparency
- Community-Based Doula (CBD) Support (Active Comparator): Pregnant patients with Medicaid insurance are screened for risk factors for low birthweight, and high-risk patients receive intensive care management. Additionally, practices receive 2 additional patient-level interventions, including: 1) Shared care of high-risk patients with Community-Based Doulas; and 2) Maternal Health Equity Education & Training sessions.
  Interventions: Other: Community-Based Doula (CBD) Support
- Data Accountability and Transparency + Community-Based Doula Support (Active Comparator): Pregnant patients with Medicaid insurance are screened for risk factors for low birthweight, and high-risk patients receive intensive care management, and practices receive all the Data Accountability and Doula Interventions described in Arms 2 and 3.
  Interventions: Other: Data Accountability and Transparency; Other: Community-Based Doula (CBD) Support

INTERVENTIONS:
Other: Data Accountability and Transparency — Collaboration with Practice Facilitators; Maternal Early Warning System; Disparities Dashboard; Racial Equity Training
  Arms: Data Accountability and Transparency; Data Accountability and Transparency + Community-Based Doula Support
Other: Community-Based Doula (CBD) Support — Community-Based Doula support for high-risk patients; Racial Equity Training
  Arms: Community-Based Doula (CBD) Support; Data Accountability and Transparency + Community-Based Doula Support

SUMMARY:
This project-also known as "Accountability for Care through Undoing Racism & Equity for Moms" or ACURE4Moms-aims to reduce Black-White maternal health disparities using multi-level interventions designed to decrease bias in prenatal care, improve care coordination, and increase social support. ACURE4Moms is a pragmatic 4-arm cluster randomized controlled trial conducted with 39 prenatal practices across North Carolina. Practices have been randomly assigned to receive either: Arm 1 (Standard Care): North Carolina Medicaid Care management for high-risk pregnancies; Arm 2 (Data Accountability and Transparency): North Carolina Medicaid Care Management + Practice-level Data Accountability interventions; Arm 3 (Community-Based Doula Support): North Carolina Medicaid Care Management + Community-Based Doula support intervention for high-risk patients during pregnancy and postpartum; or Arm 4 (Data Accountability and Transparency + Community-Based Doula Support): North Carolina Medicaid Care Management + Both Arms 2 and 3 interventions. During each practice's 2-year intervention period, the practice will initiate prenatal care for ~750-1,500 patients (up to 60,000 patients total), whose outcomes the investigators will follow and compare between arms until all these patients have reached 1-year post-delivery.

DETAILED DESCRIPTION:
Pregnancy complications are increasing in the United States, and this is worse for Black patients, who are 3-4 times more likely to die from pregnancy than White patients. Pregnancy complications and deaths cause large physical, social, and financial burdens for patients and their families. Black patients who experience higher levels of institutional racism and discrimination from healthcare providers and institutions are more likely to have pregnancy complications, such as delivering a baby with low birthweight. Low birthweight (less than 5 pounds 9 ounces) is related to many short-term and long-term health problems for both baby and mother. The study, Accountability for Care through Undoing Racism and Equity for Moms (ACURE4Moms), aims to decrease pregnancy complications for all patients, but especially for Black patients, by decreasing institutional racism and bias in healthcare and improving community-based social support during pregnancy. The primary outcome will be to decrease low birthweight deliveries among Black women. The investigators will get information about low birthweight and other pregnancy outcomes from prenatal practice electronic healthcare records. A secondary outcome will be to decrease experiences with discrimination during prenatal care among Black patients; this information will be collected from an internet survey that will be completed at 4 time points between a patient's first prenatal visit and 3 months after delivery.

To meet the study aims, the investigators will test 2 types of interventions. The first type (the "Data Accountability and Transparency interventions") will be focused on healthcare providers and their clinics. The study will improve accountability by setting up electronic Maternal Warning Systems to notify the clinics whenever a patient has a risk factor for low birthweight that needs to be treated or misses a scheduled appointment. Nurse navigators and provider champions from each clinic will make sure the clinic acts on the warning. Secondly, the study will improve transparency by showing the clinics their pregnancy-related complication data for different racial groups every 3 months through a "Disparities Dashboard." This Dashboard will show the providers any differences in pregnancy complications for people of different races in their clinic and encourage them to come up with ways to improve the quality of their care to decrease those differences. The study will hire "Practice Facilitators" to help the clinics improve their workflows and communication with patients. Finally, all the staff at the clinics will undergo interactive racial equity training to help them recognize any implicit biases they have and understand how racism affects pregnancy care for patients of color.

The second type of interventions will be focused on improving community-level support for high-risk pregnant patients. The study will do this by matching community-based doulas who are trained to provide culturally-relevant care with high-risk patients after their first prenatal appointment. The doulas will then provide support to these patients during pregnancy and up to 1 year after birth by setting up peer support groups for clients with similar due dates, attending 2 prenatal visits with them, supporting them for up to 24 hours during labor, and performing a postpartum home visit (the "Community-Based Doula Support interventions").

To test how these each of these interventions improves low birthweight alone and when combined together, the study has enrolled 39 prenatal practices across North Carolina, into 1 of 4 randomized arms: 1) No interventions; 2) Data Accountability and Transparency interventions; 3) Community-Based Doula Support interventions; or 4) Both the Data Accountability and Transparency and Community-Based Doula Support interventions. The investigators predict that up to 60,000 patients will start prenatal care at one of the 39 practices during the study.

For the patient surveys, the study plans to enroll patients who self-identify as Black or African American from each of the 39 practices, for a total of at least 2,400 survey participants. The investigators will also interview up to 250 practice staff, doulas, patients, and Practice Facilitators to understand how well the study interventions fit their needs.

The study is led by a Stakeholder Advisory Board, which includes patients of color who have had a pregnancy complication, community doulas, practice representatives, health insurance payers, a patient advocacy group, healthcare organizations, and the North Carolina Department of Public Health. The majority of members will be people of color. The Board will meet every 3 months throughout the study to advise us about patient-centered outcomes, assist with dissemination of results, and advocate for related policy change.

ELIGIBILITY:
Inclusion Criteria:

Practices:

* Have at least 180 Black patient deliver over 2 years
* Be willing to be randomized
* Be willing to adhere to the study protocol

Patient survey participants:

* Start prenatal care at one of the study clinics during study implementation
* Self-identify as Black or African American
* Able to give consent and complete surveys and interviews in English

Practice staff member participants:

* Employed as either a provider, nurse/medical assistant, or office administrator at one of the clinics in this study

Doula participants:

* Provide doula care to patients at one the clinics in this study

Exclusion Criteria:

Practices:

* Already integrated with Community-Based Doulas
* Already have an Early Warning System or Disparities Dashboard

Ages: 12 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female or transgender male
Enrollment: 30000 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Odds of delivery of low-birthweight infants among non-Hispanic Black patients in each study arm | Upon delivery
  This Primary Outcome Measure will compare the odds of delivery of low-birthweight infants (less than 2,500 grams) among non-Hispanic Black patients in each study arm as listed in the maternal delivery summary and/or neonatal electronic health record data, with the primary comparison being between the Data Accountability and Transparency + Community-Based Doula Support arm and the Standard Care arm.

SECONDARY OUTCOMES:
Odds of any discrimination during prenatal care among Black patients in each study arm | 24 weeks of gestation until delivery
  This Primary Outcome Measure will compare the odds of any perceived discrimination as measured by Discrimination in Medical Settings Scale (i.e., a score greater than or equal to 8 up to a maximum score of 35, where a higher score indicates more frequent experiences of discrimination) among Black patients in each study arm, with the primary comparison being between the Data Accountability and Transparency + Community-Based Doula Support arm and the Standard Care arm.
Odds of incidence of depression during prenatal care among Black patients in each study arm | 24 weeks of gestation until delivery
  This Secondary Outcome Measure will compare the odds of incidence of depression as measured by the Edinburgh Perinatal Depression Scale (i.e., a score greater than or equal to 10 up to a maximum score of 30, where a higher score indicates greater depressive symptoms) during prenatal care among Black patients in each study arm, with the primary comparison being between the Data Accountability and Transparency + Community-Based Doula Support arm and the Standard Care arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Tang, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill; Rachel P Urrutia, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data that documents, supports, and validates research findings will be made available after the main findings from the final research dataset have been accepted for publication. Access to databases will be available for educational, research, and non-profit purposes. All data to be shared will be stripped of any potentially identifying information. Data will be made available through a TBD data repository, in consultation with PCORI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months of publication for an unlimited period.
Access Criteria: Deidentified data will be publicly available through a TBD data repository. Research datasets may also be made available to other investigators who request access. Requests will be evaluated on a case-by-case basis by the study investigators.
  Investigators proposing to use the data will be asked to provide approval from an ethical review committee and will be asked to execute a data use/sharing agreement with UNC. Data may be shared electronically via password-protected files.
  All data sharing will abide by rules and/or policies defined by PCORI, relevant IRBs, local, state, and federal laws and regulations. Data sharing mechanisms will ensure that the rights and privacy of individuals participating in research will be protected at all times.